CLINICAL TRIAL: NCT01441154
Title: Pharmacokinetic and Pharmacodynamic Studies of Liothyronine. A Study on the Metabolic Effects of Thyroid Hormone
Brief Title: Metabolic Effects of Synthetic Thyroid Hormone for Thyroid Cancer Treatment
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110256; 11-DK-0256
Record Dates: First submitted 2011-09-24; First posted 2011-09-27 (Estimated); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Malignant Struma Ovarii; Papillary Thyroid Cancer; Hurthle Cell Thyroid Cancer; Follicular Thyroid Cancer; Tall Cell Variant Thyroid Cancer
Keywords: Hypothyroidism; Thyroid Cancer; Triiodothyronine (T3); Energy Expenditure; Thyroid Hormone
MeSH Terms: conditions — Thyroid Cancer, Papillary; Thyroid cancer, Hurthle cell; Adenocarcinoma, Follicular; Hypothyroidism; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Group 1: Adults with clinical indication for withdrawal from thyroid hormone replacement therapy in preparation for nuclear medicine imaging or therapeutic procedures with radioactive iodine

SUMMARY:
Background:

- Thyroid hormone is produced by the thyroid gland, an organ at the base of the neck. Thyroid hormone controls the body's metabolism and the function of many organs. The thyroid gland produces two forms of thyroid hormone: T4 and T3. People who have thyroid cancer are treated with thyroid hormone therapy (synthetic T4, levothyroxine), which at times needs to be stopped to allow for cancer treatments. At these times, a different form of thyroid hormone (synthetic T3, liothyronine) is used to reduce the symptoms caused by low levels of thyroid hormone. Researchers want to know more about how changes in T3 hormone affect the body and organ function.

Objectives:

- To study how changes in T3 hormone levels affect the body and organ function.

Eligibility:

- Individuals at least 18 years of age who have had most or all of their thyroid removed to treat thyroid cancer who need to stop taking their regular thyroid hormone dose in preparation for the treatment of thyroid cancer.

Design:

* The study involves a screening visit and a baseline evaluation. It also includes an 11-day inpatient hospital stay.
* Participants will be screened with a physical exam and medical history. They will also have blood tests and a neck ultrasound.
* Participants will be evaluated with a physical exam, blood tests, and the following procedures:
* Glucose tolerance test to measure blood sugar
* Tests of body fat, muscle strength, and calorie burning levels
* Imaging studies of the heart, liver, and thigh muscles
* Quality of life questionnaires
* Food preference and diet questionnaires
* After 4 weeks of treatment with T3 hormone, participants will have an 11-day inpatient hospital stay to study the effect of thyroid hormone on their metabolism. The stay will involve the same tests done in the baseline evaluation.

DETAILED DESCRIPTION:
In human adults thyroid hormone action plays a critical role in the modulation of metabolism and the function of virtually all organ/systems. The specificity of the hormonal action is ultimately the result of the interaction of the active hormone, triiodothyronine (T3), with the receptors isoforms and the co-activators and co-repressors specific for the various cells target of the hormonal action. Circulating and tissue levels of T3 are the result of the secretion of T3 and its precursor, thyroxine (T4), from the thyroid gland, the peripheral conversion of T4 into T3, and the degradation of these hormones. This complex system has only been partially studied in humans and very little is known regarding the kinetics of T3, and in particular on the correlation between circulating levels of T3 and end-organ target tissue thyroid hormone action.

The aim of this protocol is to characterize the pharmacokinetics of T3 and its biological effects at various concentrations in a cohort of thyroidectomized patients undergoing thyroid hormone replacement therapy withdrawal for the management of thyroid cancer.

Sixteen patients with a clinical indication for thyroid hormone withdrawal in preparation for 131I therapy or 123I diagnostic scan for follow-up and management of differentiated thyroid cancer will be recruited for this study. After enrollment in the study, the patients baseline characteristics will be determined during an outpatient visit while receiving levothyroxine (L-T4) therapy. The L-T4 therapy then will be suspended and substituted with an equivalent thrice daily liothyronine (L-T3) therapy for one month. Patients will be admitted to the NIH Clinical Center on the day prior to withdrawal of the T3 therapy until the diagnostic scan or the administration of radioactive iodine. During the hospitalization for this research protocol, which is expected to last eleven days, the following studies will be performed: serial blood sampling for circulating thyroid hormones to obtain pharmacokinetic parameters of L-T3, lipids, glucose and insulin, resting energy expenditure, echocardiogram, skeletal muscle strength measurement, cardiac, hepatic and skeletal muscles MRI, and quality of life and well-being questionnaires. The pharmacokinetic parameters of L-T3 will also be assessed with the first dose after the diagnostic scan or the administration of radioactive iodine.

The results obtained from this study will help in understanding the effects of thyroid hormone on metabolism, and may lead to important information on how to optimize the duration of the thyroid hormone therapy withdrawal for the treatment of thyroid cancer.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects will be adult volunteers older than age 18 who underwent total thyroidectomy for the treatment of differentiated thyroid cancer, previously undergone radioactive iodine ablation of the thyroid gland remnant, with clinical indication for withdrawal from thyroid hormone replacement therapy in preparation for nuclear medicine imaging or therapeutic procedures with radioactive iodine. The patient population will be recruited from the participants in the 77-DK-0096 natural history protocol: Studies on Thyroid Nodules and Thyroid Cancer , PI Dr.Joanna Klubo-Gwiezdzinska and from the 10-C-0102 natural history protocol: Clinical and Genetic Studies in Familial Non-Medullary Thyroid Cancer , PI Electron Kebebew.

EXCLUSION CRITERIA:

1. Significant thyroid residual greater than 5 gm as measure by ultrasound or greater than 5 percent uptake at 24 H on (123) I pre-treatment thyroid scan.
2. Renal insufficiency or estimated creatinine clearance less than or equal to 60 mL/min/1.73M(2) BSA by MDRD equation before thyroid hormone withdrawal.
3. Liver disease or ALT >2.5 times the upper laboratory reference limit.
4. Pharmacologic therapy for the treatment of psychiatric conditions.
5. History of, and/or current coronary artery disease.
6. Current history or symptoms compatible with psychosis or major depression (including history of hospitalization for depression, history of attempted suicide, history of suicidal ideation). Use of antipsychotic medications.
7. History of drug or alcohol abuse within the last year; current use of illicit drugs or alcohol abuse (CAGE>3).
8. Pregnancy (women of child-bearing potential must have a negative pregnancy test prior to inclusion) or use of hormonal contraceptives.
9. Known allergy to L-T3.
10. Current use of prescription medication or certain non-prescription medications and dietary supplements known to affect thyroid function and/or metabolism, or alter the pharmacokinetics of L-T3.
11. Inability or unwillingness to follow the low-iodine, metabolic diet or non-compliance to the L-T3 administration regimen.
12. The presence of persistent diarrhea or malabsorption syndromes that would interfere with the patient s ability to adequately absorb drugs.
13. Inability to obtain venous access for sample collection, or basal hemoglobin of less than or equal to 10 g/dL.
14. Low functional status (ECOG Performance Status > 2)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-09-20 (Actual); Primary Completion 2013-12-12 (Actual); Study Completion 2013-12-12 (Actual)

PRIMARY OUTCOMES:
1. To assess the pharmacokinetics of T3 in patients devoid of endogenous or exogenous T4 during acute L-T3 withdrawal at steady- state and after the first L-T3 dose administration | 4 weeks after stopping L-T4 thyroid hormone replacement therapy and starting L-T3 treatment
  to study T3 kinetics in thyroidectomized patients treated with liothyronine (L- T3) replacement therapy in preparation for diagnostic or therapeutic nuclear medicine procedures for the follow-up and management of differentiated thyroid cancer
2. To estimate the minimal duration of L-T3 therapy withdrawal required to achieve a serum TSH level, equal or greater than 30 uIU/mL, to assure effective 131I therapy for treatment of differentiated thyroid cancer | 4 weeks after stopping L-T4 thyroid hormone replacement therapy and starting L-T3 treatment
  to study T3 kinetics in thyroidectomized patients treated with liothyronine (L- T3) replacement therapy in preparation for diagnostic or therapeutic nuclear medicine procedures for the follow-up and management of differentiated thyroid cancer
3. To correlate clinical and biochemical parameters of thyroid hormone action, with circulating levels of T3 during L-T3 therapy withdrawal | 4 weeks after stopping L-T4 thyroid hormone replacement therapy and starting L-T3 treatment
  to study T3 kinetics in thyroidectomized patients treated with liothyronine (L- T3) replacement therapy in preparation for diagnostic or therapeutic nuclear medicine procedures for the follow-up and management of differentiated thyroid cancer

CONTACTS AND LOCATIONS:
Overall Officials: Kong Y Chen, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Yen PM. Physiological and molecular basis of thyroid hormone action. Physiol Rev. 2001 Jul;81(3):1097-142. doi: 10.1152/physrev.2001.81.3.1097. PMID 11427693
- [Background] Bianco AC, Salvatore D, Gereben B, Berry MJ, Larsen PR. Biochemistry, cellular and molecular biology, and physiological roles of the iodothyronine selenodeiodinases. Endocr Rev. 2002 Feb;23(1):38-89. doi: 10.1210/edrv.23.1.0455. PMID 11844744
- [Background] Nguyen TT, DiStefano JJ 3rd, Yamada H, Yen YM. Steady state organ distribution and metabolism of thyroxine and 3,5,3'-triiodothyronine in intestines, liver, kidneys, blood, and residual carcass of the rat in vivo. Endocrinology. 1993 Dec;133(6):2973-83. doi: 10.1210/endo.133.6.8243325.
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-DK-0256.html